CLINICAL TRIAL: NCT07333105
Title: Whole Body Vibration Versus Aerobic Training on Interleukin 6 and Endurance After Renal Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Zeinab Adel Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Zeinab-phd
Record Dates: First submitted 2026-01-01; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Whole Body Vibration; Aerobic Training; Interleukin 6; Endurance; Renal Transplantation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- whole body vibration (Experimental): In this group of the study, thirty renal transplant recipients' patients will receive the whole-body vibration for, 20 minutes 3 times per week for 12 weeks after one month post renal transplantation
  Interventions: Device: whole body vibration
- stationary bicycle (Experimental): In this group, thirty renal transplant recipients' patients will receive aerobic exercise on stationary bicycle for 20 minutes 3 times per week for 12 weeks after one month post renal transplantation
  Interventions: Device: stationary bicycle

INTERVENTIONS:
Device: whole body vibration — In a structured exercise session, subjects are instructed not to eat 2 hours prior and to wear comfortable clothing. They will rest for 10-15 minutes before starting, and will be barefoot to allow for proper vibration effects from the force platform, which induces lateral body oscillations. Before commencing, all parts of the whole-body vibration (WBV) device are checked for presence and functionality. The initial phase includes a 5-10 minute warm-up of stretching and marching. Over a 12-week period, subjects will undergo five 2-minute vibration treatments at 30 Hz, three times a week, followed by a 5-minute cool down. Participants are to stand upright with slightly flexed knees, ensuring their body alignment is maintained. Hand bars are available for those who feel insecure during the exercise.
  Arms: whole body vibration
Device: stationary bicycle — Thirty patients will undergo a supervised exercise program on a stationary bicycle for 12 weeks, exercising three times weekly. Each session will include a 5-minute warm-up (light walking), a 10-minute active phase (biking), and a 5-minute cool down (light walking). The total duration will be 20 minutes, with exercise intensity set at 60-70% of maximum heart rate, calculated using the Karvonen formula (maximum heart rate=220-Age). The walking speed will gradually increase from 60% to 70% of maximum heart rate over the course of the study.
  Arms: stationary bicycle

SUMMARY:
This study aimed to compare the effect of whole body vibration versus aerobic training on interleukin 6 and endurance after renal transplantation in patients after renal transplantation.

DETAILED DESCRIPTION:
Even after a successful renal transplantation, the renal transplant recipients (RTRs) keeps on suffering the consequences of the uremic sickness such as increased cardiovascular risk, elevated level of inflammatory cytokines (IL6), decrease work capacity and quality of life. Since biological and psychological problems are not completely solved by pharmacological treatment, physical training is able both, to improve graft function, work capacity and quality of life, and to reduce cardiovascular risk Therefore, this research aims to investigate effect of the whole-body vibration versus stationary bicycle as modes of aerobic exercises on interleukin 6 in patients and the 6-minutes walk test after renal transplantation, which may reduce the risks of cardiovascular disease, produce improvement of the biology of transplantation, increase of energetic metabolism, and allows for a better quality of life in these subtypes of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes undergone renal transplantation.
* Their age will range from 30-45 years old.
* All patients will have the same medical and nursing care.
* All the patients will receive a good explanation of treatment and measurement device.
* They will be free from any genitourinary infections.
* They will be neurologically free.

Exclusion Criteria:

* Uncooperative patients
* Instability of patient's medical condition.
* Association of another medical problem as heart disease and respiratory problems.
* Diabetic patients.
* Patients who have history of medical chronic relevant diseases.
* Patients who have acute or chronic hepatitis.
* Patients have pacemaker.
* Patients who have genitourinary infections.
* Previous history of epilepsy.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
measurement of Interleukin-6 | at baseline and 12 weeks
  Before starting the study, the following procedures will be performed. The purpose of the study will be clearly explained to each patient using simple and understandable language, and a written informed consent form will be obtained from each participant as an agreement to be included in the study. A venous blood sample (5 milliliters) will be collected from each subject in a sitting position under standardized conditions. The collected samples will be transferred into sterilized tubes containing tripotassium ethylenediaminetetraacetic acid (K3-EDTA) and heparinized tubes, which will be placed on ice and then kept at room temperature. Serum will be separated from plasma by centrifugation for 10 minutes. Interleukin-6 (IL-6) levels will be measured using the enzyme-linked immunosorbent assay (ELISA) technique with commercially available ELISA kits based on the immunoturbidimetric method. The normal reference range of interleukin-6 (IL-6) is 0-43.5 picograms per milliliter (pg/mL).

SECONDARY OUTCOMES:
assessment of functional capacity | at baseline and 12 weeks
  Subjects will be instructed to walk from end to end at the corridor of the hospital at their own pace, while attempting to cover as much distance as possible 6 min test will be evaluated before conduction of the training program and after the completion of the study Stop watch will be used for the 6-minute walk test, the test is timed with a stopwatch and the distance covered in 6 minutes walk test is used as a means to compare changes in performance capacity
assessment of endurance | at baseline and 12 weeks
  The 30-Second Chair Stand Test (30CST) evaluates leg strength and endurance in older adults as part of the Fullerton functional fitness test battery, designed to address limitations of other sit-to-stand tests. Conducted with a 17-inch folding chair, participants sit with feet shoulder-width apart and arms crossed. After a demonstration, they attempt to complete as many stands as possible in 30 seconds, maintaining proper form. Careful monitoring ensures only correctly executed stands are counted; the score reflects the total number completed, with results ranging from 0 to over 20, indicating varied fitness levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Alkahraba Hospital in Cairo, Cairo, Egypt